CLINICAL TRIAL: NCT00001955
Title: The Role of Cytokines as Inflammatory Mediators in Painful Temporomandibular Joints
Brief Title: Study of Etanercept and Celecoxib to Treat Temporomandibular Disorders (Painful Joint Conditions)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000037; 00-D-0037
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-02

CONDITIONS: Temporomandibular Joint Disorder
Keywords: Clinical Trial; Temporomandibular Joints; Celecoxib; Etanercept; Tumor Necrosis Factor; TMJ; TMD
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Etanercept; Celecoxib

INTERVENTIONS:
Drug: Etanercept
Drug: Celecoxib

SUMMARY:
This 2-part study will evaluate the effectiveness and side effects of two anti-inflammatory drugs for relieving pain and improving jaw function in patients with temporomandibular disorder (TMD). Part 1 will evaluate celecoxib (Celebrex); Part 2 will evaluate etanercept (Enbrel). The Food and Drug Administration has approved both of these drugs for treating certain forms of arthritis.

Patients between the ages of 18 and 65 years with painful jaw joint conditions may be eligible for this study. Candidates will complete several written questionnaires about their jaw condition and will undergo a medical history, complete TMD evaluation, blood and urine tests, and imaging studies of the temporomandibular joint, such as X-rays and magnetic resonance imaging. Patients will rate the quality and intensity of their pain before beginning treatment. At certain periods during the study, they will also keep a pain diary, twice a day recording the intensity and magnitude of their pain.

Part 1 - Celecoxib: Patients will be randomly assigned to receive either 1) celecoxib twice a day by mouth; 2) naproxen (a non-steroidal anti-inflammatory drug) twice a day by mouth; or 3) a placebo (inactive pill) twice a day by mouth.

Part 2 - Etanercept: Patients will be randomly assigned to receive either 1) etanercept injected under the skin or 2) saline (an inactive placebo) injected under the skin. Patients in this group will also undergo two aspirations of fluid from the jaw joint - once before treatment begins and again 6 weeks later. For this procedure, the joint is numbed with an anesthetic and then a needle is inserted into the jaw space to withdraw fluid, which will be analyzed for inflammatory processes in the joint.

All patients will have a final evaluation 6 weeks after beginning treatment, including a TMD physical examination, laboratory and X-ray tests as required. The pain diary and questionnaires will be collected at this visit.

DETAILED DESCRIPTION:
The proposed clinical trial will consist of two parallel studies. In the first part of the study, we will evaluate the analgesia and adverse effects of celecoxib, a COX-2 inhibitor in comparison to naproxen and placebo of patients with temporomandibular disorders (TMD). Celecoxib, is in oral anti-inflammatory and analgesic agent that acts by selectively inhibiting cyclooxygenase 2 (COX-2) and is not expected to cause the typical gastrointestinal, and platelet-related side effects associated with inhibition of the COX-1 enzyme. Decrease in pain, dysfunction and improvement in quality of life will be assessed at base line and after 6-week follow-up. Successful demonstration of an enhanced therapeutic effect or reduced toxicity may provide a basis for clinical use of selective COX-2 inhibitors in patients with painful TMD.

In a second group of carefully selected patients, we will evaluate the short-term effect etanercept (Enbrel) in comparison to placebo in patients who had pain and tenderness to palpation in the temporomandibular joint (TMJ osteoarthritis) of at least three month duration and who had not responded to conservative treatment. Etanercept is a biologic modifier that binds specifically to tumor necrosis factor alpha (TNF alpha). The mechanism of action of etanercept is competitive inhibition of TNF binding to cell-surface TNF receptors (TNFR), preventing TNF-mediated cellular responses by rendering TNF biologically inactive. Subjects will be randomly assigned to either etanercept or placebo administration. At baseline and at 6-week follow up individual outcomes will be assessed such as pain, mandibular range of motion along with the analysis of the sample synovial fluid level of TNF alpha. By studying the joint fluid levels of TNF alpha, we will learn more about the development of the local inflammatory process in the joint, which will help in predicting the prognosis for patients with these TM joint disorders. Positive findings will also provide clinical implications of etanercept in patients with painful TMJ osteoarthritis.

ELIGIBILITY:
Celecoxib Study:

INCLUSION CRITERIA:

Recruitment will include patients with early onset of temporomandibular disorder, whose primary diagnosis consists of anterior disc displacements with reduction as defined by the Research Diagnostic Criteria (RDC).

Subjects are required to have preauricular pain for a minimum of one month, a primary TMD diagnosis of TMJ disc displacement, and clinical and radiographic evidence of disc-displacement.

EXCLUSION CRITERIA:

Subjects who had undergone any TMJ surgery within the preceding 6 months in any active way will be excluded as will those who are taking regularly analgesic, anti-inflammatory, steroids or narcotics medications.

Further exclusion criteria will be patients who have any TMJ growth disturbances. Patients with red, hot, swollen, tendered TM joints, or those by medical history consist of infectious arthritis, crystal induced arthropathies, and musculoskeletal disorders will be excluded.

Patients will be screened for any positive history of liver or kidney dysfunctions. Patients who have known hypersensitivity to celecoxib, are allergic to sulfonamides, or have demonstrated allergic-type reactions after taking aspirin or other NSAIDs will be excluded.

Subjects that have primary psychiatric disease or score above average or higher in comparison with normative scores on Symptom Checklist (SCL-90R) will be able to participate.

Subjects with any obvious occlusal disturbances such as cross-bite, open-bite, full dentures will be disqualified.

Children under the age of 18 will be excluded from the study.

Pregnant women will not be included in the study.

Etanercept Study:

INCLUSION CRITERIA:

For the etanercept study, we will recruitment patients who are in the later stage of temporomandibular disorder, who are not responding to standard non-surgical TMD therapy (i.e., splints, physical therapy, biofeedback, trigger point injections), whose primary diagnosis consists of TMJ osteoarthritis as defined by the Research Diagnostic Criteria.

Subjects are required to have preauricular pain for a minimum of three months with clinical and radiographic evidence TMJ arthritis.

EXCLUSION CRITERIA:

Subjects who had undergone TMJ surgery within the preceding 6 months in any active way will be excluded.

Subjects that are taking regularly steroids or narcotics medications will be excluded.

Further exclusion criteria will be presence of TMJ growth disturbances. Patients with red, hot, swollen, tendered TM joints, TMJ infections or those with medical history consist of infectious arthritis, crystal induced arthropathies, and musculoskeletal disorders will be disqualified.

Patients with sepsis or with known hypersensitivity to etanercept or any of its components will be excluded from the study.

Any patients with a medical history of diabetes, congestive heart failure, or any chronic infections will be excluded.

Children under the age of 18 will not be included.

Pregnant women will not be included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1999-12; Study Completion 2004-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Allison MC, Howatson AG, Torrance CJ, Lee FD, Russell RI. Gastrointestinal damage associated with the use of nonsteroidal antiinflammatory drugs. N Engl J Med. 1992 Sep 10;327(11):749-54. doi: 10.1056/NEJM199209103271101. PMID 1501650
- [Background] Altman RD, Lozada CJ. Practice guidelines in the management of osteoarthritis. Osteoarthritis Cartilage. 1998 May;6 Suppl A:22-4. doi: 10.1016/s1063-4584(98)80007-1. PMID 9743815
- [Background] Arend WP, Dayer JM. Cytokines and cytokine inhibitors or antagonists in rheumatoid arthritis. Arthritis Rheum. 1990 Mar;33(3):305-15. doi: 10.1002/art.1780330302. PMID 2180403